CLINICAL TRIAL: NCT06969885
Title: The Effect of Virtual Reality Glasses Applied Before Coronary Angiography on Patients' Stress Levels, Muscle Tension, and Certain Physiological Parameters
Brief Title: Effect of Virtual Reality Glasses on Stress, Muscle Tension, and Physiological Parameters Before Angiography
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yuksek Ihtisas University (Other)
Responsible Party: Principal Investigator, Aylin GÜÇLÜ DEMİREL, Assistant Professor (PhD), Yuksek Ihtisas University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2024/215
Record Dates: First submitted 2025-04-17; First posted 2025-05-14 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Coronary Angiography (CAG)
Keywords: Coronary Angiography; Virtual Reality Glasses; Stress; Muscle Tension; Physiological Parameters

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Other): No intervention will be made to the patients outside of the hospital routine, and approximately 10 minutes before the procedure, the Physiological Parameters Monitoring Form, Distress Thermometer and VAS will be applied again and the data collection process will be completed.
  Interventions: Behavioral: Standard application
- Experimental Group (Experimental): In the preoperative period, approximately 1 hour before the procedure, a video will be watched for 15 minutes with virtual reality glasses. Approximately 10 minutes before the procedure, the patients will be administered the Physiological Parameters Monitoring Form, Distress Thermometer and VAS, and the data collection process will be completed.
  Interventions: Behavioral: Intervention application with virtual reality glasses

INTERVENTIONS:
Behavioral: Intervention application with virtual reality glasses — In the preoperative period, approximately 1 hour before the procedure, a video will be watched for 15 minutes with virtual reality glasses. Approximately 10 minutes before the procedure, the patients will be administered the Physiological Parameters Monitoring Form, Distress Thermometer and VAS, and the data collection process will be completed.
  Arms: Experimental Group
Behavioral: Standard application — No intervention will be made to the patients outside of the hospital routine, and approximately 10 minutes before the procedure, the Physiological Parameters Monitoring Form, Distress Thermometer and VAS will be applied again and the data collection process will be completed.
  Arms: Control Group

SUMMARY:
Today, cardiovascular diseases are the leading cause of morbidity and mortality worldwide. Coronary angiography (CAG), a commonly used invasive procedure for diagnosing coronary artery disease, may trigger fear, stress, and anxiety in patients due to its invasive nature, lack of information, uncertainty, and the possibility of receiving a life-threatening diagnosis.These emotional responses activate stress mechanisms, leading to catecholamine release, increased heart rate, blood pressure, respiration, sweating, and muscle tension. Elevated stress can also cause lactic acid accumulation, increased oxygen demand, and muscular contraction, potentially resulting in coronary artery spasms or arrhythmias, and increasing procedural risks. Therefore, reducing stress before CAG is crucial to improving procedural outcomes and patient recovery.

To address preoperative anxiety and stress, both pharmacologic and non-pharmacologic interventions are used. Among the non-pharmacologic options, virtual reality (VR) has emerged as an effective method to distract and calm patients, reducing anxiety, stress, and pain. Studies in various patient populations suggest VR glasses can be beneficial in managing psychological distress. However, no study has been found in the literature evaluating the effect of VR on stress-induced muscle tension in patients undergoing CAG. This gap highlights the potential contribution of this study to current knowledge.

This study aims to investigate the effect of using VR glasses before coronary angiography on patients' stress levels, muscle tension, and selected physiological parameters.

DETAILED DESCRIPTION:
Study Hypotheses:

H0: There is no difference in preoperative stress, muscle tension, or physiological parameters.

H1: There is a difference in preoperative stress levels. H2: There is a difference in preoperative muscle tension. H3: There is a difference in certain physiological parameters preoperatively. H4: There is a relationship between stress, muscle tension, and physiological parameters preoperatively.

ELIGIBILITY:
Inclusion Criteria: - 18-65 years of age,

* Scheduled to undergo CAG,
* American Society of Anesthesiologists (ASA) score I or II,
* Turkish-speaking patients will be included.

Exclusion Criteria: Patients with nausea,

* with dizziness,
* with headache,
* with any known psychiatric disease and mental perception problem,
* pregnant,
* with a history of epilepsy,
* with vision, hearing and perception problems,
* with closed space phobia,
* with a history of dizziness, nausea, etc. due to previous virtual reality use will not be included in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Distress Thermometer | Preoperative period
  It is a Likert-type scale with scores from 0 (no stress) to 10 (extreme stress) developed by Roth et al. (1998) to determine psychological distress in cancer patients. In the short and easy-to-understand scale, patients can easily mark their own stress levels within the specified ranges on the thermometer. The Turkish validity-reliability study of the Distress Thermometer was conducted by Özalp et al. (2007) . In their study, Özmen and Gürsoy (2021) concluded that the distress thermometer can be used as a valid and reliable measurement tool to measure the stress experienced by patients who will undergo surgery. With this scale, the stress levels of the patients in the last week and at the time of evaluation will be evaluated.
Assessment of Muscle Tension | Preoperative period
  Measuring patients' symptomatic experiences through questionnaires or self-reports is the gold standard method for assessing the presence and severity of a mental disorder. In a study conducted by Sainsbury and Gibson (1954) on symptoms reported by anxious, stressed patients, "feeling of tension" was mostly defined as "feeling of tension in the muscles," "muscle stiffness," "cramping," and "body discomfort" line with this information, the 10-point Visual Analogy Scale (VAS) will be used to assess muscle tension resulting from stress in patients before the CAG procedure, and patients will be asked to rate their feelings of tension in the muscles, stiffness in the muscles, cramping in any muscle, and inability to relax their body using this scale. This scale is 10 centimeters (cm) long and includes numbers from 0 to 10. The values marked by the patient between 0-10 cm on the scale will be ta
Physiological Parameters Monitoring Form | Preoperative period
  This form includes questions about patients' systolic and diastolic blood pressure
Physiological Parameters Monitoring Form | Preoperative period
  This form includes question about patients' pulse
Physiological Parameters Monitoring Form | Preoperative period
  This form includes question about patients' respiratory rate
Physiological Parameters Monitoring Form | Preoperative period
  This form includes question about patients' oxygen saturation.

SECONDARY OUTCOMES:
Distress Thermometer | Approximately 10 minutes before the procedure, patients
  The patients were reapplied approximately 10 minutes before the procedure to measure their stress levels.
Assessment of Muscle Tension | About 10 minutes before entering the process
  Patients will be asked to rate whether they feel tension in their muscles, a feeling of stiffness in their muscles, a feeling of cramping in any muscle, or an inability to relax their body.
Physiological Parameters Monitoring Form | About 10 minutes before entering the process
  Approximately 10 minutes before the procedure, patients are asked questions about their systolic and diastolic blood pressure
Physiological Parameters Monitoring Form | About 10 minutes before entering the process
  Approximately 10 minutes before the procedure, patients are asked question about pulse
Physiological Parameters Monitoring Form | About 10 minutes before entering the process
  Approximately 10 minutes before the procedure, patients are asked question respiratory rate
Physiological Parameters Monitoring Form | About 10 minutes before entering the process
  Approximately 10 minutes before the procedure, patients are asked question about oxygen saturation.

CONTACTS AND LOCATIONS:
Locations (1):
- Yüksek İhtisas University, Ankara, Çankaya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No